CLINICAL TRIAL: NCT01589848
Title: Study on Von Willebrand Disease and Hemophilia in Cuenca, Ecuador
Acronym: VWD
Status: Completed | Type: Observational
Sponsor: Universidad del Azuay (Other)
Responsible Party: Principal Investigator, Jaime M. Moreno A., M.D., M.S., F.A.C.P., Jaime M. Moreno A, M.D., M.S., F.A.C.P., Universidad del Azuay
Other Study IDs: 001; UAzuay (Other Grant/Funding Number: Universidad del Azuay, Cuenca, Ecuador)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Von Willebrand Disease; Hemophilia A; Hemophilia B
Keywords: vWD
MeSH Terms: conditions — von Willebrand Diseases; Hemophilia A; Hemophilia B

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- von Willebrand women: Referred women who may have von Willebrand Disease

SUMMARY:
1. Hypothesis

   a. There are patients with von Willebrand Disease in Cuenca.
2. Primary question

   a. How many women referred with a history of bleeding may have von Willebrand disease?
3. Secondary

   1. Associations between the bleeding score and initial laboratory studies
   2. What are the differences on subgroups of enrolled patients with the bleeding score?
4. Ancillary

   1. What is the clinical and socio-economic status of women with von Willebrand Disease in Cuenca?
   2. What is the clinical and socio-economic status of patients with Hemophilia in Cuenca?

DETAILED DESCRIPTION:
The incidence of hemophilia A is 1 in 10,000 and the one of hemophilia B is 1 in 30,000 live born males. As the most frequent coagulopathy in the world, von Willebrand disease (vWD) can affect 1 in 1000 children of both genders. The prevalence of vWD is 1-2% and it may be as high as 5-15% among women with menorrhagia. So vWD can be present in 1 of every 100 to 500 individuals.

A world survey published that Ecuador, with a population of 14,790,608 people, has 238 patients with hemophilia, 45 people with von Willebrand disease (vWD) and 13 patients with other bleeding disorders including rare factor deficiencies and platelet disorders.

The Ecuadorian census of 2010 indicates that Cuenca district (canton) has 505,585 inhabitants. According to a local reference, Cuenca has no reports of vWD and it has registered 20-40 patients with hemophilia A and B. However Cuenca may host approximately 10,000 people with vWD because it affects both males and females. One plausible explanation for this lag is that the diagnostic suspicions of vWD had not been proven because of the lack of a special coagulation laboratory in Cuenca that would allow professionals to make a positive diagnosis.

This is the first clinical, demographic and socio-economic study of patients registered with hemophilia and of Cuenca women with possible vWD who are referred from dentists and physicians from public and private health centers. The instruments will be validated surveys and screening coagulation studies.

As far as we know Ecuador has not published studies on coagulopathies. Our aim is to initiate a process to eventually reach the goal to offer adequate diagnostic and therapeutic interventions to human victims of these diseases, within a program of service, teaching and research.

ELIGIBILITY:
Inclusion Criteria:

* Subjects living at urban and rural parishes from Cuenca district.
* Subjects referred from professionals of public and private health services, who have filled the initial hemorrhage survey.
* Must be referred women who sign the informed consent form.
* Patients who answer the standardized bleeding score questionnaire (BS).
* Patients who answer the quality of life questionnaire (SF-12).
* Patients who answer the socio-economic survey.
* Patients who accept to provide a venous blood sample for the initial laboratory tests.

Exclusion Criteria:

* Women with organic or hormonal bleeding etiologies.
* Patients taking medicines which may affect the coagulation cascade or the number or function of platelets.
* Those women who otherwise do not comply with the inclusion criteria.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Target population: all women from Cuenca district with a hemorrhage history.
  Accessible population: Those women referred from professionals with an initial hemorrhage history, who comply with the inclusion criteria and who sign the informed consert form.
  Sample population: First comers referred with a hemorrhage history until fulfilling the projected sample size. This non-probabilistic purposive sample will be used because it has been reported that it could represent the target population.
  *2010 Ecuadorian census: 131.163 women ages 18 to 50 years, at Cuenca district.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bleeding Score (BS) | 1 week
  As an adequate bleeding history is fundamental, the Condensed MCMDM-1 Bleeding Questionnaire will be used. Its bleeding score (BS) has a sensitivity of 100%, specificity 87%, positive predictive value 0.2 and negative predictive value 1.0. There was a signifficant difference of BS between the subtypes of vWD: with type 3 >>type 2 >>type 1 vWD (Anova P <0.001).
  AS the BS is an index of ordinal values, medians and the Mann-Whitney non-parametric ranksum test will be used, to study the bleeding score (BS) differences among subgroups of enrolled women.

SECONDARY OUTCOMES:
Associations among BS and female subgroup characteristics and initial laboratory tests. | 1 week
  As bleeding may tend to associate in subjects, i.e. epistaxis and menorrhagia, a logistic (log-linear) model will be used. As bleeding can also ocur independently, symptoms will be coded for an adjusted covariate analysis.
  To study the relationships among the BS and the quantitative laboratory results, the BS will be divided in quintiles, and an adjusted multiple regression model will be used. Likelihood ratios (LR) for values of BS, with a prevalence of 5% and ROC curves will be applied. According to Tosetto et.al. laboratory data will be expressed in categorical and quantitative scales.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime M. Moreno A., M.D., M.S., Principal Investigator — Universidad del Azuay (UAzuay); Jacinto Guillen G., Eng., M.S., Study Chair — Universidad del Azuay (UAzuay); Rodrigo Cueva M., Econ., M.S., Study Director — Universidad del Azuay (UAzuay)
Locations (2):
- Ecuador (2):
  - UAzuay, Cuenca, Azuay
  - Universidad del Azuay (UDA), Cuenca, Azuay